CLINICAL TRIAL: NCT00924287
Title: Phase I/II Study of Metastatic Cancer That Expresses Her-2 Using Lymphodepleting Conditioning Followed by Infusion of Anti-Her-2 Gene Engineered Lymphocytes
Brief Title: Gene Therapy Using Anti-Her-2 Cells to Treat Metastatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated after the first patient treated on study died as a result of the treatment.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090041; 09-C-0041; NCT00805987 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2012-02-14 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Cancer
Keywords: Metastatic Cancer; Tumor Regression; Immunotherapy; Safety; Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — Receptors, Chimeric Antigen; Automobiles; aldesleukin; Interleukin-2; Cyclophosphamide; fludarabine; fludarabine phosphate; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metastatic Cancer (Experimental): Cancer that has invaded other parts of the body
  Interventions: Drug: in vitro tumor reactive, chimeric T cell receptor (CAR ) gene-transduced PBL plus IV aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna

INTERVENTIONS:
Drug: in vitro tumor reactive, chimeric T cell receptor (CAR ) gene-transduced PBL plus IV aldesleukin — 720,000 IU/kg every 8 hours for a maximum of 15 doses
  Other Names: Proleukin; IL-2; Interleukin-2
Drug: Cyclophosphamide — 60 mg/kg/day x 2 days intravenously (IV) in 250 ml 5% dextrose in water (D5W) with mesna 15 mg/kg/day x 2 days over 1 hour
  Other Names: Cytoxan; Neosar; Endoxan; Procytox; Revimmune
Drug: Fludarabine — 25 mg/m^2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara
Drug: Mesna — 3 mg/kg/hour intravenously diluted in a suitable diluent over 23 hours after each cyclophosphamide dose.
  Other Names: Mesnex; Uromitexan

SUMMARY:
Background:

* Human epidermal growth factor receptor-2 (Her-2) is a gene found in both normal cells and cancer cells. Extra copies of the gene (overexpression) can cause too many Her-2 proteins (receptors) to appear on the cell surface and cause tumors to grow.
* An experimental procedure developed for treating patients with cancer uses blood cells found in their tumors or bloodstream. The cells are genetically modified using the anti-Her-2 gene and a type of virus. The modified cells (anti-Her-2 cells) are grown in the laboratory and then given back to the patient to try to decrease the size of the tumors. This is called gene therapy.

Objectives:

* To determine whether advanced cancers that overexpress Her-2 can be treated effectively with lymphocytes (white blood cells) that have been genetically engineered to contain an anti-Her-2 protein.

Eligibility:

* Patients 18 years of age and older with metastatic cancer (cancer that has spread beyond the original site) and for whom standard treatments are not effective.
* Patient's tumor overexpresses Her-2.

Design:

* Workup with scans, x-rays and other tests.
* Leukapheresis to obtain cells for preparing the anti-Her-2 cells for later infusion.
* 1 week of chemotherapy to prepare the immune system for receiving the anti-Her-2 cells.
* Infusion of anti-Her-2 cells, followed by interleukin-2 (IL-2) treatment. The cells are given as an infusion through a vein. IL-2 is given as a 15-minute infusion through a vein every 8 hours for a maximum of 15 doses.
* Periodic follow-up clinic visits after hospital discharge for physical examination, review of treatment side effects, laboratory tests and scans every 1 to 6 months.

DETAILED DESCRIPTION:
Background:

* We have constructed a single retroviral vector that contains a chimeric T cell receptor (CAR) that recognizes the Her-2 tumor antigen, which can be used to mediate genetic transfer of this CAR with high efficiency (greater than 30%) without the need to perform any selection.
* In co-cultures with Her-2 positive tumors, anti-Her-2 CAR transduced T cells secreted significant amount of interferon-gamma (IFN-gamma) (Her-2 high specificity).

Objectives:

Primary objectives:

* To evaluate the safety of the administration of anti-Her-2 -CAR engineered peripheral blood lymphocytes in patients receiving the non-myeloablative conditioning regimen and aldesleukin.
* Determine if the administration of anti-Her-2 -CAR engineered peripheral blood lymphocytes and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer that expresses the Her-2 antigen.

Secondary objective:

- Determine the in vivo survival of CAR gene-engineered cells.

Eligibility:

Patients who are 18 years of age or older must have

* metastatic cancer whose tumors express the Her-2 antigen;
* previously received and have been a non-responder to or recurred after standard care for metastatic disease;

Patients may not have:

- contraindications for high dose aldesleukin administration.

Design:

* Peripheral blood mononuclear cell (PBMC) obtained by leukapheresis (approximately 5 times 10^9 cells) will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of approximately 10^8 to 5 times 10^8 cells to retroviral vector supernatant containing the anti-Her-2 CAR genes .
* Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous (IV) infusion of ex vivo tumor reactive, CAR genetransduced PBMC plus IV aldesleukin (720,000 IU/kg q8h for a maximum of 15 doses).
* Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment. If the patient has stable disease (SD) or tumor shrinkage, repeat complete evaluations will be performed every 1-3 months. After the first year, patients continuing to respond will continue to be followed with this evaluation every 3-4 months until off study criteria are met.
* The study will be conducted using a Phase I/II optimal design. The protocol will proceed in a phase 1 dose escalation design, with three cohorts. Should a single patient experience a dose limiting toxicity (DLT) at a particular dose level, three more patients would be treated at that dose to confirm that no greater than 1/6 patients have a DLT prior to proceeding to the next higher level. If a level with 2 or more DLTs in 3-6 patients has been identified, three additional patients will be accrued at the next-lowest dose, for a total of 6, in order to further characterize the safety of the maximum tolerated dose prior to starting the phase II portion. If a dose limiting toxicity occurs in the first cohort, that cohort will be expanded to 6 patients. If 2 DLTs are encountered in this cohort, the study will be terminated.
* Once the maximum tolerated dose (MTD) has been determined, the study then would proceed to the phase II portion. Patients will be entered into two cohorts based on histology: cohort 1 will include patients with metastatic breast cancer, and cohort 2 will include patients with other types of metastatic cancer that express Her-2.
* For each of the 2 strata evaluated, the study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. For each of these two arms of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.
* The objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, and anti-Her-2 CAR-gene engineered lymphocytes is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% partial response (PR) + complete response (CR) rate (p1=0.20).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Metastatic cancer that expresses Her-2 at greater than or equal to 2+ and assessed by immunohistochemistry (IHC) in the clinical laboratory improvement amendment (CLIA) approved test in the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI), National Institutes of Health (NIH).
  2. Patients must have previously received systemic standard care (or effective salvage chemotherapy regimens) for metastatic disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred. Subjects with estrogen receptor-positive or progesterone receptor-positive breast cancer must have progressed on or not be a candidate for anti-estrogens or aromatase inhibitors and all breast cancer patients must have progressed on or not be a candidate for an anthracycline-containing regimen and a taxane-containing regimen.
  3. Patients with breast cancer must have previously received trastuzumab. Patients will not continue to receive trastuzumab during the trial period.
  4. Greater than or equal to 18 years of age.
  5. Willing to sign a durable power of attorney
  6. Able to understand and sign the Informed Consent Document
  7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  8. Life expectancy of greater than three months.
  9. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the preparative regimen.
  10. Serology:

      1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
      2. Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcriptase polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
      3. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
  11. Hematology:

      1. Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
      2. White blood cell (WBC) (> 3000/mm^3).
      3. Platelet count greater than 100,000/mm^3.
      4. Hemoglobin greater than 8.0 g/dl.
  12. Chemistry:

      1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
      2. Serum creatinine less than or equal to 1.6 mg/dl.
      3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  13. Left ventricular ejection fraction (LVEF) greater than or equal to 50%.
  14. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
  15. Patients who have previously received anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) antibody therapy must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
2. Active systemic infections; coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system; myocardial infarction; cardiac arrhythmias; obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent Systemic steroid therapy
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of coronary revascularization or ischemic symptoms
8. Documented forced expiratory volume in 1 second (FEV1) less than or equal to 60% predicted tested in patients with:

   1. A prolonged history of cigarette smoking (20 pack/year of smoking within the past 2 years).
   2. Symptoms of respiratory dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Sakaguchi K, Robbins PF, Rivoltini L, Yannelli JR, Appella E, Rosenberg SA. Identification of the immunodominant peptides of the MART-1 human melanoma antigen recognized by the majority of HLA-A2-restricted tumor infiltrating lymphocytes. J Exp Med. 1994 Jul 1;180(1):347-52. doi: 10.1084/jem.180.1.347. PMID 7516411
- [Background] Dudley ME, Wunderlich J, Nishimura MI, Yu D, Yang JC, Topalian SL, Schwartzentruber DJ, Hwu P, Marincola FM, Sherry R, Leitman SF, Rosenberg SA. Adoptive transfer of cloned melanoma-reactive T lymphocytes for the treatment of patients with metastatic melanoma. J Immunother. 2001 Jul-Aug;24(4):363-73. doi: 10.1097/00002371-200107000-00012. PMID 11565838
- [Background] Dudley ME, Wunderlich JR, Yang JC, Hwu P, Schwartzentruber DJ, Topalian SL, Sherry RM, Marincola FM, Leitman SF, Seipp CA, Rogers-Freezer L, Morton KE, Nahvi A, Mavroukakis SA, White DE, Rosenberg SA. A phase I study of nonmyeloablative chemotherapy and adoptive transfer of autologous tumor antigen-specific T lymphocytes in patients with metastatic melanoma. J Immunother. 2002 May-Jun;25(3):243-51. doi: 10.1097/01.CJI.0000016820.36510.89. PMID 12000866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was accrued to this study.
Period: Overall Study
Arm/Group | Metastatic Cancer
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Metastatic Cancer
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Clinical Tumor Regression Response
Description: Response Evaluation Criteria in Solid Tumors (RECIST) are used to determine objective clinical response. Complete Rresponse (CR) is the disappearance of all target lesions, partial response (PR) is at least a 30% decrease in the target lesions, progressive disease (PD) is at least a 20% increase in the target lesions or appearance of one or more new lesions, and stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: 12 days
Arm/Group | Metastatic Cancer
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 12 days
Measure: Number; unit: Participants
Arm/Group | Metastatic Cancer
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Number of Participants With In Vivo Survival of Transfused Cells
Description: In-vivo survival of infused cells is determined by analysis of the sequence of the variable region of the T cell receptor or flow cytometry (FACS).
Time Frame: 12 days
Measure: Number; unit: Participants
Arm/Group | Metastatic Cancer
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 12 days
Arm/Group | Metastatic Cancer
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic Cancer (N=1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic Cancer (N=1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (2)
Leukocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (2)
Fibrinogen decreased (Blood and lymphatic system disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Metabolism and nutrition disorders) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Bilirubin increased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (2)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Low urine output (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated after the first patient on study died as a result of the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No